CLINICAL TRIAL: NCT03717883
Title: Endogenous Molecule Profiling in Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: ADPKD Alterations in Hepatic Transporter Function
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-2984; 5R35GM122576-02 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: ADPKD; Autosomal Dominant Polycystic Kidney Disease; Renal Disease
Keywords: hepatic transporters
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples used for potential studies will not be labeled with personal identifiers and will be stored for up to 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects
- Subjects with ADPKD

SUMMARY:
This is a single center, comparative cohort study to investigate alterations in hepatic transporter function in subjects with autosomal dominant polycystic kidney disease (ADPKD) compared to healthy subjects and subjects with non-ADPKD renal disease. Eligible subjects will be 18-65 years of age and of any race/ethnicity and gender.

DETAILED DESCRIPTION:
ADPKD is a relatively common genetic disease affecting about 1 out of every 1000 people worldwide. Progression of ADPKD is characterized by the proliferation of fluid-filled kidney cysts. Development of these cysts is progressive and can lead to end-stage renal disease and ultimately, renal failure in many patients. The most common extra-renal complication of ADPKD is the formation of liver cysts, which can vary from minor to extensive. Hepatic cysts can develop from medium-sized bile ducts and complications (i.e., cyst rupture, infection, obstruction of bile ducts, and compromised portal venous flow) can arise from increasing cystic burden. Previous studies have shown that elevated levels of endogenous molecules such as bile acids in ADPKD may indicate altered transporter function. Other endogenous molecules such as coproporphyrin (CP) I and III may be used as probes to assess hepatic transporter function.

The objective of this study is to investigate and quantify ADPKD-associated alterations in endogenous molecule profiles (e.g., bile acids, CP) relative to subjects with non-ADPKD renal disease and healthy individuals, and to investigate specific hepatic transporter polymorphisms that may be related to the alterations. This is important because subjects with ADPKD may be predisposed to adverse reactions associated with some medications that require hepatic transporters for excretion.

Potential study participants will be pre-screened over the phone and then scheduled for a 2-hour study visit. All urine samples within the 2-hour interval will be collected from all participants along with clinical, physical and questionnaire data. Fasting blood samples will be collected at time 0 and 120 min.

ELIGIBILITY:
Inclusion Criteria (all subjects):

* Provide signed and dated informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 18 to 65
* Negative quantitative human chorionic gonadotropin (hCG) blood test (for women of child-bearing age only)

For healthy subjects:

* Normal liver functions tests (LFTs) as defined by the University of North Carolina (UNC) hospital laboratory reference range [aspartate aminotransferase (AST)14-38 U/L, alanine aminotransferase (ALT) 15-48 U/L, alkaline phosphatase 38-126 U/L]
* Normal clinical laboratory results including kidney function (serum creatinine) and lipid panel as reviewed by the study physician

For subjects with ADPKD:

* Man or woman between the ages of 18 and 65 with documented ADPKD

For subjects with non-ADPKD renal disease:

* Man or woman between the ages of 18 and 65 with documented non-ADPKD renal disease as determined by the study physician

Exclusion Criteria:

All Participants:

* Donation of blood within the last 30 days
* Diagnosis of human immunodeficiency virus (HIV) and/or untreated hepatitis C virus (HCV)
* History of significant alcohol abuse and/or illicit drug use
* More than 1 glass of wine or 2 beers (or equivalent in % alcohol) per day during the 48 hours prior to study and/or screening visit
* Inability to fast for 8 hours prior to study and screening sample collection
* Women who are pregnant, trying to become pregnant, or breastfeeding
* Current or recent (within 30 days) use of bile acid sequestrants, bile acid derivatives (i.e. ursodiol) or fibric acid derivatives
* History of diabetes or taking blood glucose lowering treatments
* Radiologic imaging consistent with cirrhosis and portal hypertension
* Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dL, total bilirubin > 1.5 mg/dL, or prothrombin time (PT)/international normalized ratio (INR) > 1.3 times normal at screening, or history or presence of ascites, encephalopathy, or bleeding from esophageal varices
* Estimated glomerular filtration rate (GFR)< 15 mL/min per 1.73 m2, or on dialysis, at screening
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications (including inhaled) within 14 days of study visit. Corticosteroids with minimal systemic absorption (for example topical) and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease provided the dose has been stable for ≥4 weeks and is not expected to change during the course of the study.
* Primary, secondary or extra-hepatic malignancy
* BMI > 35 kg/m2 at screening
* Inability or unwillingness to give informed consent or abide by the study protocol
* History or other evidence of illness, any gastrointestinal surgery (e.g., gall bladder removal), or any other conditions or drug therapies that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, gall bladder disease, active gastrointestinal conditions or taking drugs known to interfere with bile acid synthesis or metabolism or the metabolism/transport of other drugs)

Healthy Subjects:

* Taking concomitant medications, both prescription and non-prescription (including herbal products and over-the-counter medications), other than oral contraceptives and multivitamins (women stabilized on hormonal methods of birth control will be allowed to participate)
* History or other evidence of liver, gall bladder, or intestinal disease in the opinion of the study investigators
* BMI > 35 kg/m2 at screening.

Subjects with non-ADPKD renal disease:

* ADPKD
* Proteinuria of ≥3 grams per day of protein into the urine; or on a single spot urine collection, the presence of ≥2 grams of protein per gram of urine creatinine (i.e., excluding patients with nephrotic-range proteinuria)
* Diabetic nephropathy patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy vs. ADPKD vs. non-ADPKD renal disease subjects
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Difference in serum coproporphyrin I and III concentrations | 2 hours
  nmol

SECONDARY OUTCOMES:
Difference in serum and urine bile acid profiles | 2 hours
  nmol
Difference in renal clearance of coproporphyrin I and III | 2 hours
  mL/min

CONTACTS AND LOCATIONS:
Overall Officials: Vimal Derebail, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Kim Brouwer, PharmD, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Igarashi P, Somlo S. Genetics and pathogenesis of polycystic kidney disease. J Am Soc Nephrol. 2002 Sep;13(9):2384-98. doi: 10.1097/01.asn.0000028643.17901.42. No abstract available. PMID 12191984
- [Background] Boucher C, Sandford R. Autosomal dominant polycystic kidney disease (ADPKD, MIM 173900, PKD1 and PKD2 genes, protein products known as polycystin-1 and polycystin-2). Eur J Hum Genet. 2004 May;12(5):347-54. doi: 10.1038/sj.ejhg.5201162. PMID 14872199
- [Background] Cnossen WR, Drenth JP. Polycystic liver disease: an overview of pathogenesis, clinical manifestations and management. Orphanet J Rare Dis. 2014 May 1;9:69. doi: 10.1186/1750-1172-9-69. PMID 24886261
- [Background] Salam M, Keeffe EB. Liver cysts associated with polycystic kidney disease: role of Tc-99m hepatobiliary imaging. Clin Nucl Med. 1989 Nov;14(11):803-7. doi: 10.1097/00003072-198911000-00003. PMID 2598550
- [Background] Hofmann AF. The continuing importance of bile acids in liver and intestinal disease. Arch Intern Med. 1999 Dec 13-27;159(22):2647-58. doi: 10.1001/archinte.159.22.2647. PMID 10597755
- [Background] Zollner G, Fickert P, Silbert D, Fuchsbichler A, Marschall HU, Zatloukal K, Denk H, Trauner M. Adaptive changes in hepatobiliary transporter expression in primary biliary cirrhosis. J Hepatol. 2003 Jun;38(6):717-27. doi: 10.1016/s0168-8278(03)00096-5. PMID 12763363
- [Background] Kullak-Ublick GA, Stieger B, Meier PJ. Enterohepatic bile salt transporters in normal physiology and liver disease. Gastroenterology. 2004 Jan;126(1):322-42. doi: 10.1053/j.gastro.2003.06.005. PMID 14699511
- [Background] Munoz-Garrido P, Marin JJ, Perugorria MJ, Urribarri AD, Erice O, Saez E, Uriz M, Sarvide S, Portu A, Concepcion AR, Romero MR, Monte MJ, Santos-Laso A, Hijona E, Jimenez-Aguero R, Marzioni M, Beuers U, Masyuk TV, LaRusso NF, Prieto J, Bujanda L, Drenth JP, Banales JM. Ursodeoxycholic acid inhibits hepatic cystogenesis in experimental models of polycystic liver disease. J Hepatol. 2015 Oct;63(4):952-61. doi: 10.1016/j.jhep.2015.05.023. Epub 2015 Jun 1. PMID 26044126
- [Background] Shen H, Dai J, Liu T, Cheng Y, Chen W, Freeden C, Zhang Y, Humphreys WG, Marathe P, Lai Y. Coproporphyrins I and III as Functional Markers of OATP1B Activity: In Vitro and In Vivo Evaluation in Preclinical Species. J Pharmacol Exp Ther. 2016 May;357(2):382-93. doi: 10.1124/jpet.116.232066. Epub 2016 Feb 23. PMID 26907622
- [Background] Gilibili RR, Chatterjee S, Bagul P, Mosure KW, Murali BV, Mariappan TT, Mandlekar S, Lai Y. Coproporphyrin-I: A Fluorescent, Endogenous Optimal Probe Substrate for ABCC2 (MRP2) Suitable for Vesicle-Based MRP2 Inhibition Assay. Drug Metab Dispos. 2017 Jun;45(6):604-611. doi: 10.1124/dmd.116.074740. Epub 2017 Mar 21. PMID 28325716
- [Background] Devuyst O, Chapman AB, Gansevoort RT, Higashihara E, Perrone RD, Torres VE, Blais JD, Zhou W, Ouyang J, Czerwiec FS. Urine Osmolality, Response to Tolvaptan, and Outcome in Autosomal Dominant Polycystic Kidney Disease: Results from the TEMPO 3:4 Trial. J Am Soc Nephrol. 2017 May;28(5):1592-1602. doi: 10.1681/ASN.2016040448. Epub 2016 Dec 5. PMID 27920153
- [Background] Watkins PB, Lewis JH, Kaplowitz N, Alpers DH, Blais JD, Smotzer DM, Krasa H, Ouyang J, Torres VE, Czerwiec FS, Zimmer CA. Clinical Pattern of Tolvaptan-Associated Liver Injury in Subjects with Autosomal Dominant Polycystic Kidney Disease: Analysis of Clinical Trials Database. Drug Saf. 2015 Nov;38(11):1103-13. doi: 10.1007/s40264-015-0327-3. PMID 26188764
- [Background] Lai Y, Mandlekar S, Shen H, Holenarsipur VK, Langish R, Rajanna P, Murugesan S, Gaud N, Selvam S, Date O, Cheng Y, Shipkova P, Dai J, Humphreys WG, Marathe P. Coproporphyrins in Plasma and Urine Can Be Appropriate Clinical Biomarkers to Recapitulate Drug-Drug Interactions Mediated by Organic Anion Transporting Polypeptide Inhibition. J Pharmacol Exp Ther. 2016 Sep;358(3):397-404. doi: 10.1124/jpet.116.234914. Epub 2016 Jun 17. PMID 27317801
- [Background] Brock WJ, Beaudoin JJ, Slizgi JR, Su M, Jia W, Roth SE, Brouwer KLR. Bile Acids as Potential Biomarkers to Assess Liver Impairment in Polycystic Kidney Disease. Int J Toxicol. 2018 Mar/Apr;37(2):144-154. doi: 10.1177/1091581818760746. PMID 29587557
- [Background] Ferslew BC, Xie G, Johnston CK, Su M, Stewart PW, Jia W, Brouwer KL, Barritt AS 4th. Altered Bile Acid Metabolome in Patients with Nonalcoholic Steatohepatitis. Dig Dis Sci. 2015 Nov;60(11):3318-28. doi: 10.1007/s10620-015-3776-8. Epub 2015 Jul 3. PMID 26138654
- [Background] Gurka MJ, Coffey CS, Gurka KK. Internal pilots for observational studies. Biom J. 2010 Oct;52(5):590-603. doi: 10.1002/bimj.201000050. PMID 20857422
- [Background] Jennison C, Turnbull BW. Adaptive sample size modification in clinical trials: start small then ask for more? Stat Med. 2015 Dec 20;34(29):3793-810. doi: 10.1002/sim.6575. Epub 2015 Jul 14. PMID 26172385
- [Background] Coffey CS, Muller KE. Properties of internal pilots with the univariate approach to repeated measures. Stat Med. 2003 Aug 15;22(15):2469-85. doi: 10.1002/sim.1466. PMID 12872303
- [Background] Denne JS. Sample size recalculation using conditional power. Stat Med. 2001 Sep 15-30;20(17-18):2645-60. doi: 10.1002/sim.734. PMID 11523074